CLINICAL TRIAL: NCT03364049
Title: Phase 1b Open-label Study of MK-7162 in Combination With Pembrolizumab (MK-3475) +/- Other Therapies in Participants With Advanced Solid Tumors
Brief Title: Study of MK-7162 in Combination With Pembrolizumab (MK-3475) in Adult Participants With Advanced Solid Tumors (MK-7162-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7162-002; 2017-000418-49 (EudraCT Number); MK-7162-002 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Solid Neoplasms
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MK-7162 25 mg +Pembrolizumab (Pembro) (Experimental): Participants receive MK-7162 25 mg via oral tablets once daily (QD) throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 25 mg orally QD PLUS pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (every 3 weeks [Q3W]).
  Interventions: Drug: MK-7162; Biological: Pembrolizumab
- MK-7162 50 mg + Pembro (Experimental): Participants receive MK-7162 50 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-71625 50 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
  Interventions: Drug: MK-7162; Biological: Pembrolizumab
- MK-7162 100 mg + Pembro (Experimental): Participants receive MK-7162 100 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 100 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
  Interventions: Drug: MK-7162; Biological: Pembrolizumab
- MK-7162 200 mg + Pembro (Experimental): Participants receive MK-7162 200 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 200 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
  Interventions: Drug: MK-7162; Biological: Pembrolizumab

INTERVENTIONS:
Drug: MK-7162 — oral tablets
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; Keytruda

SUMMARY:
The purposes of this study are to determine the safety and tolerability of MK-7162 when administered in combination with pembrolizumab (MK-3475) and to establish a preliminary recommended Phase 2 dose (RP2D) of MK-7162 when administered in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically- or cytologically-confirmed advanced/metastatic solid tumor by pathology report and have received, or been intolerant to, or been ineligible for all treatment known to confer clinical benefit. Participants with solid tumors of any type are eligible for enrollment.
* Has stage III or stage IV disease that is not surgically resectable.
* Has measurable disease by RECIST 1.1 criteria as assessed by the local site investigator/radiology.
* Has 1 or more discrete malignant lesions that are amenable to ≥2 separate biopsies guided by one of the following modalities: visual inspection, ultrasound guidance, or cross sectional image guidance (computed tomography/magnetic resonance imaging [CT/MRI]).
* Has an evaluable baseline tumor sample to submit for analysis.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrates adequate organ function.
* If male, must agree to use contraception and refrain from donating sperm during the treatment period and for ≥120 days after last dose of study treatment.
* If female, is not pregnant or breastfeeding, and if a woman of childbearing potential (WOCCBP), agrees to use contraception during the treatment period and for ≥120 days after last dose of study treatment.

Exclusion Criteria:

* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. (Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers.)
* Has a known active central nervous system metastasis and/or carcinomatous meningitis.
* Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody/components of the study treatment(s).
* Has an active autoimmune disease that has required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy.
* Has a history of vasculitis.
* Has an active infection requiring systemic therapy.
* Has symptomatic ascites or pleural effusion.
* Has interstitial lung disease that has required oral or intravenous glucocorticoids to assist with management.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years. (Note: Participants who have had a stem cell transplant >5 years ago are eligible as long as there are no symptoms of graft-versus-host disease [GVHD].)
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has known active Hepatitis B or known active Hepatitis C virus infection.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Has not fully recovered from any effects of major surgery without significant detectable infection.
* Has received prior systemic anti-cancer therapy including investigational agents or has used an investigational device within 28 days prior to the first dose of study treatment. (Notes: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Prior exposure to immunotherapeutics is allowed, including programmed cell death-1 (PD-1) and programmed cell death-ligand 1 (PD-L1) inhibitors, provided the participant did not experience ≥Grade 3 drug-related toxicity on monotherapy with a PD-1 or PD-L1 inhibitor.
* Has been previously treated with an Indoleamine-2,3-dioxygenase-1 (IDO1) inhibitor (e.g., epacadostat, BMS-986205)
* Has received prior radiotherapy within 2 weeks of start of study treatment.
* Is receiving a monoamine oxidase inhibitor (MAOI) or any drug which has significant MAOI activity (e.g., meperidine, linezolid, methylene blue) within the 21 days before screening, or has a history of Serotonin Syndrome after receiving serotonergic drugs.
* Is expected to require any non-protocol antineoplastic therapy while on study.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy in excess of replacement doses (the equivalent of prednisone ≤10 mg/day is acceptable), or on any other form of immunosuppressive medication.
* Has received a live-virus vaccine within 30 days prior to first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- United States (3):
  - UCLA Medical Center ( Site 0002), Santa Monica, California
  - START Midwest ( Site 0007), Grand Rapids, Michigan
  - Laura and Isaac Perlmutter Cancer Center ( Site 0001), New York, New York
- Princess Margaret Hospital.. ( Site 0130), Toronto, Ontario, Canada
- Chaim Sheba Medical Center. ( Site 0301), Ramat Gan, Israel
- Severance Hospital Yonsei University Health System ( Site 0103), Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a screening period to determine eligibility. 41 participants were screened for this study and 33 were randomized.
Groups:
- MK-7162 25 mg + Pembrolizumab (Pembro): Cycle 1: Participants receive MK-7162 25 mg via oral tablets once daily (QD) throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 25 mg orally QD PLUS pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle (every 3 weeks [Q3W]).
Period: Overall Study
Arm/Group | MK-7162 25 mg + Pembrolizumab (Pembro) | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Started | 6 | 6 | 6 | 15
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 15
Not completed — Death | 6 | 4 | 5 | 14
Not completed — In survival phase status at study closure. Participant transferred to pembrolizumab extension study | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- MK-7162 25 mg + Pembro: Participants receive MK-7162 25 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 25 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
- Total: Total of all reporting groups
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro | Total
Number analyzed (Participants) | 6 | 6 | 6 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (14.5) | 56.0 (14.2) | 61.7 (9.9) | 59.6 (12.8) | 59.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 8 | 20
  Male | 2 | 2 | 2 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 5 | 6 | 6 | 12 | 29
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 2 | 3
  White | 5 | 5 | 3 | 7 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-limiting Toxicities (DLTs) as Assessed Using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 by the Investigator
Description: The following events, if considered drug related by the investigator, are considered a DLT: Grade 4 nonhematologic toxicity; Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia; Grade 4 thrombocytopenia of any duration; Grade 3 thrombocytopenia associated with bleeding; Nonhematologic Adverse Events (AE) ≥Grade 3 with exceptions; Grade 3 or Grade 4 non-hematologic laboratory values if requires medical intervention, leads to hospitalization, persists for >1 week, or results in a Drug-induced Liver Injury with exceptions; Grade 3 of 4 febrile neutropenia; Treatment-related toxicities that lead to discontinuation of study treatment during Cycles 1 or 2; Prolonged delay (>2 weeks) in initiating Cycles 2 or 3 due to treatment-related toxicity; Missing >25% of MK-7162 doses as a result of treatment-related AE during Cycles 1 or 2; Grade 5 toxicity.
Time Frame: Cycle 1 and Cycle 2 (Up to 6 weeks)
Population: All participants who received at least one dose of study treatment and were observed for safety for 21 days after the first dose of assigned treatment or experienced a DLT prior to 21 days after the first dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 6 | 15
Participants | 0 | 0 | 0 | 5

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.
Time Frame: Up to Approximately 27 Months
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 6 | 15
Participants | 6 | 6 | 6 | 15

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to Approximately 26 Months
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 6 | 15
Participants | 0 | 0 | 1 | 4

4. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) From 0-8 Hours of MK-7261 Alone and in Combination With Pembrolizumab
Description: Blood samples were collected at designated time points for determining the AUC₀-₈ of MK-7162 in plasma when administered alone and in combination with pembrolizumab.
Time Frame: Pre-dose and at 1, 2, 4, and 8 hours post-dose on Cycle 1, Days 1 & 15; and Cycle 3, Day 1
Population: All participants who were compliant with the study procedures and have available data from at least one treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 5 | 14
hr*nM
  Day 1, Cycle 1: MK-7162 alone | 4400 (36.5) | 8640 (29.9) | 20700 (32.6) | 31700 (44.4)
  Day 15, Cycle 1: MK-7162 alone: number analyzed (Participants) | 5 | 5 | 5 | 11
  Day 15, Cycle 1: MK-7162 alone | 10300 (37.3) | 19200 (90.7) | 47300 (87.8) | 118000 (93.5)
  Day 1, Cycle 3: MK-7162 + Pembrolizumab: number analyzed (Participants) | 4 | 3 | 3 | 5
  Day 1, Cycle 3: MK-7162 + Pembrolizumab | 12200 (27.7) | 20900 (101.2) | 36100 (117.8) | 10700 (98.4)

5. Secondary Outcome: Minimum Plasma Concentration (Cmin) of MK-7162
Description: Blood samples were obtained at designated time points to determine the Cmin of MK-7162 in plasma.
Time Frame: Pre-dose and at 1, 2, 4, and 8 hours post-dose on Cycle 1, Day 14
Population: All participants who were compliant with the study procedures and have available plasma data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 5 | 5 | 5 | 11
nM | 1070 (73.1) | 1260 (219.9) | 3390 (130.3) | 13800 (177.3)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-7162 When Administered Alone and in Combination With Pembrolizumab
Description: Blood samples were collected at designated time points to determine the Cmax of MK-7162 in plasma when administered alone and in combination with pembrolizumab.
Time Frame: Pre-dose and at 1, 2, 4, and 8 hours post-dose on Cycle 1, Days 1 and 15 and Cycle 3, Day 1
Population: All participants who were compliant with the study procedures and have available data from at least one treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 6 | 14
nM
  Day 1 Cycle 1: MK-7162 alone: number analyzed (Participants) | 6 | 6 | 5 | 14
  Day 1 Cycle 1: MK-7162 alone | 902 (48.0) | 1750 (27.8) | 4420 (28.2) | 6550 (48.6)
  Day15 Cycle 1: MK-7162 Alone: number analyzed (Participants) | 5 | 5 | 5 | 11
  Day15 Cycle 1: MK-7162 Alone | 1940 (38.3) | 3560 (64.1) | 8910 (84.5) | 20600 (77.0)
  Day 1 Cycle 3: MK-7162+ Pembrolizumab: number analyzed (Participants) | 4 | 4 | 3 | 6
  Day 1 Cycle 3: MK-7162+ Pembrolizumab | 2140 (52.2) | 3120 (96.2) | 6110 (100.9) | 17800 (77.9)

7. Secondary Outcome: Kynurenine (KYN) Biomarker Plasma Concentration
Description: MK-7162 is a selective inhibitor of Indoleamine-2,3-dioxygenase-1 (IDO1) activity which, in turn, reduces the conversion of TRP to KYN. Venous blood samples were collected after an overnight fast for measurement of plasma levels of KYN as a pharmacodynamic biomarker of IDO1 inhibition.
Time Frame: Cycle 1 Days 1 & 15: predose, 1, 2, 4 & 8 hours postdose; Cycle 2 Day 1: predose; Cycle 3 Day 1: predose, 1, 2, 4 & 8 hours postdose; Cycle 3 Day 15: predose
Population: All participants who were compliant with the study procedures and have available data from at least one treatment
Measure: Mean (Full Range); unit: μmol/L
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 6 | 15
μmol/L
  Cycle 1 Day 1, Predose | 1.9 [1.2 to 2.7] | 1.5 [1.2 to 2.2] | 2.3 [1.4 to 3.4] | 1.7 [0.5 to 2.5]
  Cycle 1 Day 1, 1 Hour (hr) Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day 1, 1 Hour (hr) Postdose | 1.9 [1.1 to 2.5] | 1.5 [1.1 to 1.8] | 2.2 [1.4 to 3.2] | 1.5 [0.5 to 2.2]
  Cycle 1 Day 1, 2 Hr Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day 1, 2 Hr Postdose | 2.0 [1.2 to 2.7] | 1.5 [1.1 to 2.1] | 2.2 [1.4 to 3.2] | 1.5 [0.6 to 2.5]
  Cycle 1 Day 1, 4 Hr Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day 1, 4 Hr Postdose | 2.0 [1.5 to 2.6] | 1.5 [1.2 to 1.9] | 2.1 [1.3 to 3.0] | 1.5 [0.6 to 2.4]
  Cycle 1 Day1, 8 Hr Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day1, 8 Hr Postdose | 1.8 [1.1 to 2.6] | 1.4 [0.9 to 1.9] | 2.0 [1.1 to 2.7] | 1.4 [0.6 to 2.6]
  Cycle 1 Day 15, Predose: number analyzed (Participants) | 5 | 6 | 6 | 12
  Cycle 1 Day 15, Predose | 1.6 [1.0 to 2.3] | 1.2 [0.8 to 1.5] | 1.3 [0.4 to 2.3] | 1.0 [0.6 to 2.2]
  Cycle 1 Day 15, 1 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 12
  Cycle 1 Day 15, 1 Hr Postdose | 1.7 [1.0 to 2.6] | 1.2 [0.9 to 1.4] | 1.3 [0.3 to 2.3] | 1.0 [0.6 to 2.3]
  Cycle 1 Day 15, 2 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 14
  Cycle 1 Day 15, 2 Hr Postdose | 1.8 [1.3 to 2.6] | 1.2 [0.8 to 1.5] | 1.3 [0.4 to 2.2] | 1.0 [0.6 to 2.1]
  Cycle 1 Day 15, 4 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 14
  Cycle 1 Day 15, 4 Hr Postdose | 1.8 [1.3 to 2.8] | 1.2 [1.0 to 1.6] | 1.3 [0.4 to 2.1] | 1.1 [0.6 to 2.4]
  Cycle 1 Day 15, 8 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 14
  Cycle 1 Day 15, 8 Hr Postdose | 1.7 [1.0 to 2.3] | 1.1 [0.9 to 1.4] | 1.2 [0.2 to 2.1] | 1.0 [0.6 to 2.2]
  Cycle 2 Day 1, Predose: number analyzed (Participants) | 2 | 1 | 6 | 4
  Cycle 2 Day 1, Predose | 2.1 [1.2 to 2.1] | 1.2 [1.2 to 1.2] | 0.6 [0.6 to 0.7] | 1.0 [0.6 to 1.7]
  Cycle 3 Day 1, Predose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, Predose | 1.8 [1.1 to 2.5] | 1.6 [1.1 to 1.9] | 1.4 [0.4 to 2.3] | 1.1 [0.4 to 2.3]
  Cycle 3 Day 1, 1 Hr Postdose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, 1 Hr Postdose | 1.8 [1.0 to 2.4] | 1.6 [1.3 to 2.0] | 1.3 [0.4 to 2.3] | 1.1 [0.4 to 2.2]
  Cycle 3 Day 1, 2 Hr Postdose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, 2 Hr Postdose | 2.0 [1.0 to 2.8] | 1.6 [1.2 to 1.8] | 1.4 [0.1 to 2.3] | 1.1 [0.4 to 2.4]
  Cycle 3 Day 1, 4 Hr Postdose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, 4 Hr Postdose | 2.0 [1.2 to 2.9] | 1.6 [1.3 to 1.9] | 1.4 [0.4 to 2.5] | 1.1 [0.3 to 2.3]
  Cycle 3 Day 1, 8 Hr Postdose: number analyzed (Participants) | 4 | 5 | 3 | 9
  Cycle 3 Day 1, 8 Hr Postdose | 1.8 [1.0 to 2.6] | 1.6 [1.2 to 1.9] | 1.4 [0.5 to 2.4] | 1.1 [0.2 to 2.3]
  Cycle 3 Day 15, PreDose: number analyzed (Participants) | 6 | 6 | 2 | 7
  Cycle 3 Day 15, PreDose | 2.0 [0.9 to 3.0] | 2.2 [1.3 to 4.1] | 1.5 [1.4 to 1.6] | 0.9 [0.5 to 1.9]

8. Secondary Outcome: Tryptophan (TRP) Biomarker Plasma Concentration
Description: MK-7162 is a selective inhibitor of Indoleamine-2,3-dioxygenase-1 (IDO1) activity which, in turn, reduces the conversion of TRP to KYN. Venous blood samples were collected at designated time points after an overnight fast for measurement of plasma levels of TRP as a pharmacodynamic biomarker of IDO1 inhibition.
Time Frame: as for outcome 7
Population: All participants who were compliant with the study procedures and have available data from at least one treatment
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 6 | 15
mg/dL
  Cycle 1 Day1, Predose | 0.7 [0.5 to 1.0] | 0.8 [0.5 to 1.1] | 0.7 [0.3 to 1.1] | 0.7 [0.3 to 1.4]
  Cycle 1 Day 1, 1 Hr Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day 1, 1 Hr Postdose | 0.7 [0.5 to 0.9] | 0.8 [0.5 to 1.2] | 0.6 [0.3 to 0.8] | 0.6 [0.3 to 1.4]
  Cycle 1 Day 1, 2 Hr Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day 1, 2 Hr Postdose | 0.8 [0.5 to 1.1] | 0.9 [0.4 to 1.3] | 0.7 [0.4 to 0.9] | 0.7 [0.2 to 1.6]
  Cycle 1 Day 1, 4 Hr Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day 1, 4 Hr Postdose | 0.9 [0.6 to 1.1] | 0.9 [0.4 to 1.2] | 0.7 [0.4 to 1.0] | 0.8 [0.5 to 1.7]
  Cycle 1 Day 1, 8 Hr Postdose: number analyzed (Participants) | 6 | 6 | 5 | 15
  Cycle 1 Day 1, 8 Hr Postdose | 0.9 [0.6 to 1.2] | 0.9 [0.4 to 1.7] | 0.8 [0.4 to 1.0] | 0.8 [0.4 to 1.4]
  Cycle 1 Day 15, Predose: number analyzed (Participants) | 5 | 6 | 6 | 12
  Cycle 1 Day 15, Predose | 0.8 [0.6 to 0.9] | 0.8 [0.6 to 0.9] | 0.6 [0.2 to 1.2] | 0.7 [0.3 to 1.6]
  Cycle 1 Day 15, 1 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 12
  Cycle 1 Day 15, 1 Hr Postdose | 0.9 [0.6 to 1.0] | 0.7 [0.5 to 0.9] | 0.6 [0.2 to 1.0] | 0.7 [0.3 to 1.4]
  Cycle 1 Day 15, 2 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 14
  Cycle 1 Day 15, 2 Hr Postdose | 0.9 [0.8 to 1.0] | 0.8 [0.5 to 1.1] | 0.6 [0.3 to 1.0] | 0.6 [0.3 to 1.2]
  Cycle 1 Day 15, 4 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 14
  Cycle 1 Day 15, 4 Hr Postdose | 1.0 [0.6 to 1.1] | 0.8 [0.5 to 1.0] | 0.7 [0.4 to 1.1] | 0.7 [0.4 to 1.6]
  Cycle 1 Day 15,8 Hr Postdose: number analyzed (Participants) | 5 | 6 | 6 | 14
  Cycle 1 Day 15,8 Hr Postdose | 1.0 [0.8 to 1.1] | 0.8 [0.5 to 1.0] | 0.7 [0.2 to 1.2] | 0.7 [0.3 to 1.7]
  Cycle 2 Day 1, Predose: number analyzed (Participants) | 2 | 1 | 2 | 4
  Cycle 2 Day 1, Predose | 0.8 [0.8 to 0.9] | 0.6 [0.6 to 0.6] | 0.7 [0.3 to 1.0] | 0.6 [0.4 to 1.0]
  Cycle 3 Day 1, Predose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, Predose | 0.8 [0.5 to 0.9] | 0.7 [0.6 to 0.8] | 0.5 [0.2 to 0.8] | 0.7 [0.2 to 1.2]
  Cycle 3 Day 1, 1 Hr Postdose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, 1 Hr Postdose | 0.8 [0.7 to 0.8] | 0.7 [0.5 to 0.9] | 0.5 [0.2 to 0.7] | 0.7 [0.3 to 1.4]
  Cycle 3 Day 1, 2 Hr Postdose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, 2 Hr Postdose | 0.9 [0.8 to 1.1] | 0.8 [0.7 to 1.0] | 0.6 [0.2 to 0.9] | 0.7 [0.4 to 1.4]
  Cycle 3 Day 1, 4 Hr Postdose: number analyzed (Participants) | 4 | 5 | 3 | 10
  Cycle 3 Day 1, 4 Hr Postdose | 0.9 [0.8 to 1.0] | 0.8 [0.6 to 0.9] | 0.6 [0.2 to 0.8] | 0.8 [0.4 to 1.4]
  Cyle 3 Day 1, 8 Hr Postdose: number analyzed (Participants) | 4 | 5 | 6 | 9
  Cyle 3 Day 1, 8 Hr Postdose | 0.9 [0.4 to 1.2] | 0.7 [0.5 to 0.8] | 0.6 [0.3 to 0.9] | 0.8 [0.4 to 1.4]
  Cycle 3 Day 15, Predose: number analyzed (Participants) | 6 | 6 | 2 | 7
  Cycle 3 Day 15, Predose | 0.8 [0.5 to 1.0] | 0.6 [0.3 to 0.7] | 0.6 [0.4 to 0.8] | 0.6 [0.3 to 1.2]

9. Secondary Outcome: Objective Response Rate (ORR) Based on Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by the Investigator
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 as assessed by the Investigator. The percentage of participants who experience a CR or PR based on RECIST 1.1 will be presented.
Time Frame: Up to approximately 28 months
Population: All participants with a baseline scan that demonstrated measurable disease by the investigator's assessment, and who were administered at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 6 | 6 | 6 | 15
Percentage of Participants | 0.0 [0.0 to 45.9] | 16.7 [0.4 to 64.1] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 21.8]

10. Secondary Outcome: Overall Response Based on Immune Response Evaluation Criteria (iRECIST) In Solid Tumors
Description: Participants with PD by RECIST 1.1 as determined by investigator underwent confirmatory imaging to classify the disease as confirmed progressive disease (iCPD), unconfirmed progressive disease [iUPD]), stable disease (iSD), partial response (iPR) or complete response (iCR). iCPD definition: Worsening of target lesions (increase in the sum of diameters of ≥5 mm); Any significant growth in non-target lesions, Appearance of new lesions, increase in new lesion sum of diameters by ≥5 mm; Visible growth of new non-target lesions; or appearance of new factor that would have triggered PD by RECIST 1.1. Responses are classified as iSD or iPR (depending on the sum of diameters of the target lesions), or iCR if all lesions resolve. iUPD overall response is defined as none of the progression-confirming factors identified in iCPD occurs AND The target lesion sum of diameters (initial target lesions) remains above the initial PD threshold (by RECIST 1.1)
Time Frame: Up to approximately 28 months
Population: All participants who had follow up tumor imaging subsequent to initial progressive disease per RECIST 1.1 by investigator assessment
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-7162 25 mg + Pembro | MK-7162 50 mg + Pembro | MK-7162 100 mg + Pembro | MK-7162 200 mg + Pembro
Number analyzed (Participants) | 5 | 5 | 3 | 12
Percentage of Participants
  iCR | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 26.5]
  iPR | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 26.5]
  iSD | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 26.5]
  iUPD | 80.0 [28.4 to 99.5] | 60.0 [14.7 to 94.7] | 100.0 [29.2 to 100.0] | 75.0 [42.8 to 94.5]
  iCPD | 20.0 [0.5 to 71.6] | 40.0 [5.3 to 85.3] | 0.0 [0.0 to 70.8] | 25.0 [5.5 to 57.2]

ADVERSE EVENTS:
Time Frame: Up to approximately 27 months
Description: The safety analysis population includes all participants who received at least one dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study treatment are excluded as AEs.
Groups:
- MK-7162 25mg + Pembro: Participants receive MK-7162 25 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 25 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
- MK-7162 50mg + Pembro: Participants receive MK-7162 50 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 50 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
- MK-7162 100mg + Pembro: Participants receive MK-7162 100 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 100 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
- MK-7162 200mg + Pembro: Participants receive MK-7162 200 mg via oral tablets QD throughout the 3-week cycle. Cycles 2 through 36: Participants receive MK-7162 200 mg orally QD PLUS pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle Q3W
Arm/Group | MK-7162 25mg + Pembro | MK-7162 50mg + Pembro | MK-7162 100mg + Pembro | MK-7162 200mg + Pembro
All-Cause Mortality (participants affected / at risk) | 6/6 | 4/6 | 5/6 | 14/15
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/6 | 3/6 | 5/15
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7162 25mg + Pembro (N=6) | MK-7162 50mg + Pembro (N=6) | MK-7162 100mg + Pembro (N=6) | MK-7162 200mg + Pembro (N=15)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Afferent loop syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-7162 25mg + Pembro (N=6) | MK-7162 50mg + Pembro (N=6) | MK-7162 100mg + Pembro (N=6) | MK-7162 200mg + Pembro (N=15)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (6) | 2 (2) | 3 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (3) | 3 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3) | 3 (3) | 9 (9)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (3) | 1 (4) | 2 (5) | 4 (6)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (2) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 0 (0) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship should reflect significant contribution to the design and conduct of the trial, performance or interpretation of the analysis, and/or writing of the manuscript. All named authors must be able to defend the trial results and conclusions. Merck funding of a trial will be acknowledged in publications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT03364049/Prot_SAP_000.pdf